CLINICAL TRIAL: NCT04749901
Title: Symptoms of Post-traumatic Stress in Adult Drug-resistant Epilepsies: Incidence and Influence on Cognitive Control Capacities and on Seizure Control
Brief Title: Symptoms of Post-traumatic Stress in Adult Drug-resistant Epilepsies
Acronym: SPIRALE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossible to pursue the study
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-42; ID-RCB (Other: 2020-A01829-30)
Record Dates: First submitted 2021-01-14; First posted 2021-02-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with epilepsy (Other)
  Interventions: Other: Psycho-emotional and semiological measures
- Patients with PTSD (Other)
  Interventions: Other: Psycho-emotional and semiological measures
- Patients with type 1 diabetes (Other)
  Interventions: Other: Psycho-emotional and semiological measures
- Patients with a heart rhythm disorder (Other)
  Interventions: Other: Psycho-emotional and semiological measures

INTERVENTIONS:
Other: Psycho-emotional and semiological measures — Surveys, interviews and measures
  Other Names: Cognitive measures; Physiological measurements; Qualitative measures

SUMMARY:
Epilepsy is a neurological disease that can cause many comorbid psychiatric disorders, among them: generalized anxiety disorder and depression. Many studies suggest a temporal relationship between exposure to a traumatic event and the development of epilepsy. The objective of this research is to study the symptoms of post-traumatic stress disorder (PTS) in patients with epilepsy, and their relation to anxiety and depression in these patients. The investigators also wish to study how such symptoms may be associated with the subjective semiological manifestations of epileptic seizures. In addition, it has been shown that patients with epilepsy are able, from the identification of different warning signs, to anticipate their vulnerability to having an epileptic seizure allowing them to set up different types. strategies to control them. The investigators also wish to study the cognitive processes involved in this control and the influence of PTS symptoms, in particular hypervigilance on this behavior.

The investigators propose a protocol using different types of measures: emotional, cognitive and physiological in order to answer our questions. In addition to patients with epilepsy, two groups of patients will be included: a group of patients with another chronic non-neurological disease to compare the prevalence of PTS symptoms and a group of patients with post-traumatic stress disorder ( PTSD) to compare with patients with epilepsy, cognitive and physiological measures.

Finally, the results of this study should allow to develop tools for assessing PTS symptoms in epilepsy and to develop specific management approaches

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 50 years old;
* Native French speaker;
* Level of education higher than the 3rd school level;
* Certain diagnosis of the pathology of the experimental group with which he will be associated, more precisely:
* Group of patients with epilepsy [Group E]: definite diagnosis of drug-resistant epilepsy (epileptic seizures persist despite the administration of daily treatment) established by a specialist physician.
* Group of patients with a heart rhythm disorder [Group C]: definite diagnosis of one of the following disorders: Atrial Fibrillation (AF); Syncope and Bouveret's disease established by a specialist.
* Group of patients with T1 diabetes mellitus [Group D]: definite diagnosis of type 1 diabetes established by a specialist doctor.
* Group of patients with PTSD [Group T]: definite diagnosis of PTSD established by a specialist doctor.
* Person having given his non-objection

Exclusion Criteria:

* Pregnancy;
* Breastfeeding women;
* Severe cognitive impairment
* Addiction to alcohol or drugs (including drugs other than those related to epilepsy or the chronic disease from which the patient has);
* Other neurological and / or psychiatric disorders than CNEP or epilepsy except anxiety and depressive disorders;
* Adults under guardianship or under judicial protection
* People deprived of their liberty
* Inability to read French.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Baseline
  Beck Anxiety inventory (0-63), higher values mean worse outcome
Depression | Baseline
  Beck Anxiety inventory (0-21), higher values mean worse outcome
Number of patients with PTSD | Baseline
  Post-traumatic stress disorder
Emotion regulation | Baseline
  The difficulties in emotion regulation scale,(0-180), higher values mean better outcome
Quality of life of the patient | Baseline
  Medical Outcome Study and 36-item Short Form Health Survey (0-60),higher values mean worse outcome
Seizures control | Baseline
  Seizure control scale (0-85), higher values mean better outcome
Seizures control (heart rythm) | Baseline
  HRSC
PTSD | Baseline
  PTSD-E (0-100), higher values mean worse outcome
Emotionnal control of diabete | Baseline
  DID-C (Diabete insulino-dependant-Control) (elaborated for the study) (0-150), higher values mean worse outcome
Emotionnal control of diabete and PTSD | Baseline
  DID-PTSD (Diabete insulino-dependant-Posttraumatic Stress Disorder) (elaborated for the study) (0-185), higher values mean worse outcome
Skin conductance | Baseline
  BIOPAC SCL (EDA 100C)
Eyes movements | Baseline
  EyeLink 1000 (SR Research)
Heart rythm variability | Baseline
  BIOPAC ECG (EL250)
Attentional and executive control | Baseline
  Attentional and executive control task in the context of hypervigilance (elaborated for the study) (0-180), higher values mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No